CLINICAL TRIAL: NCT00892411
Title: Prognostic Value of Measures of Central Hypersensitivity in Patients With Low Back Pain
Brief Title: Prognostic Value of Measures of the Central Hypersensitivity in Patients With Acute Low Back Pain
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: KEK 103/08
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Pain Measurement; Low Back Pain
Keywords: Neuroplasticity; Prognosis
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All study participants: Patients With Acute Low Back Pain

SUMMARY:
Background. Patients with chronic low back pain display hyperexcitability of the central nervous system (central hypersensitivity). Such hypersensitivity may occur in the acute phase and represent a risk factor for the development of chronic pain.

Objective. To determine the prognostic value of central hypersensitivity for the development of chronic low back pain.

Design. Prospective cohort study.

Setting. Primary care.

Patients. 140 individuals with acute low back pain and no history of chronic pain.

Outcomes. Primary prognostic variable will be the pain tolerance threshold at the second toe (the pressure intensity at which a further increase in pressure is deemed intolerable). Exploratory secondary prognostic variables are measures of mechanisms related to central hypersensitivity: stimulus-specific hypersensitivity (pressure, electrical, heat and cold stimulation); tissue-specific hypersensitivity (skin vs. muscle stimulation); localized vs. widespread hypersensitivity; spinal cord modulation (electrophysiological measures of hypersensitivity and changes in receptive fields); modulation at brain level (descending modulation of nociceptive input and cortical plasticity). Clinical primary outcome will be the occurrence of chronic low back pain at follow-up.

Main analysis. The investigators will use least square logistic regression models to determine the association of central hypersensitivity with prognosis.

Relevance. An understanding of the prognostic value of central hypersensitivity may allow an early stratification for treatment of individuals at risk of developing chronic low back pain. Subgroups of patients may be selected for clinical trials on novel pharmacological approaches for the prevention and treatment of central hypersensitivity.

DETAILED DESCRIPTION:
Background

Prolonged afferent nociceptive input induces an increase in the excitability of central sensory neurons and plasticity changes that cause hyperexcitability of the central nervous system (central hypersensitivity. The hyperexcitable central nervous system amplifies the nociceptive signal, thereby producing an exaggerated pain response even in the presence of limited tissue damage.

Using quantitative sensory tests, central hypersensitivity has been detected in different chronic musculoskeletal pain syndromes. Patients with chronic low back pain display increased pain sensitivity and enlargement of the areas of referred pain after stimulation of tissues around and distant from the site of pain (i.e. the leg or the thumb), suggesting that widespread central hypersensitivity is associated with this condition. Functional reorganization of the cortex has been detected in different pain conditions, including low back pain. Using equal levels of sensory stimulation in patients and pain-free controls, patients with chronic low back pain showed more extensive patterns of neuronal activation in pain-related cortical areas.

An investigation on patients after a whiplash injury found that those patients with persistent moderate or severe symptoms at 6 months had displayed, soon after injury, widespread hypersensitivity. Therefore, central hypersensitivity may be an indicator of poor prognosis. An acute peripheral lesion may induce plasticity changes leading to central hypersensitivity in a subset of individuals. Such a hypersensitivity would facilitate the transition from acute to chronic pain and disability. This hypothesis has been investigated using a limited number of tests only in a limited number of individuals with whiplash injury, but not in any other condition.

Objective

To determine the prognostic value of different measures of mechanisms of central hypersensitivity in patients with acute low back pain.

Methods

140 consecutive Patients with acute low back pain, referred by general practice, will be studied prospectively. Primary prognostic variable will be the pain tolerance threshold at the second toe (the pressure intensity at which a further increase in pressure is deemed intolerable). Exploratory secondary prognostic variables are measures of mechanisms related to central hypersensitivity: stimulus-specific hypersensitivity (pressure, electrical, heat and cold stimulation); tissue-specific hypersensitivity (skin vs. muscle stimulation); localized vs. widespread hypersensitivity; spinal cord modulation (electrophysiological measures of hypersensitivity and changes in receptive fields); modulation at brain level (descending modulation of nociceptive input and cortical plasticity). Clinical primary outcome will be the occurrence of chronic low back pain at follow-up. The investigators will use least square logistic regression models to determine the association of central hypersensitivity with prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Acute low back pain < 6 weeks
* Age 18-80

Exclusion Criteria

* History of chronic low back pain
* Radicular pain
* Pregnancy
* Breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute low back pain referred from primary care.
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2009-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Presence or absence of chronic low back pain | 6 months after the acute episode

SECONDARY OUTCOMES:
Mechanisms of central hypersensitivity | During the acute episode of low back pain

CONTACTS AND LOCATIONS:
Overall Officials: Michele Curatolo, MD, PhD, Study Director — Dep. of Anesthesiology and Pain Therapy, Bern University Hospital; Monika Müller, MD, PhD, Principal Investigator — Dep. of Anesthesiology and Pain Therapy, Bern University Hospital
Locations (1):
- Dep. of Anesthesiology and Pain Therapy, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Derived] Vuilleumier PH, Arguissain FG, Biurrun Manresa JA, Neziri AY, Nirkko AC, Andersen OK, Arendt-Nielsen L, Curatolo M. Psychophysical and Electrophysiological Evidence for Enhanced Pain Facilitation and Unaltered Pain Inhibition in Acute Low Back Pain Patients. J Pain. 2017 Nov;18(11):1313-1323. doi: 10.1016/j.jpain.2017.05.008. Epub 2017 Jun 20. PMID 28645867